CLINICAL TRIAL: NCT04561349
Title: Effects of Task Oriented Training on Walking in Children With Cerebral Palsy
Brief Title: Effects of TOT on Walking in Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00242 Madiha Tariq
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Walking; Task oriented training; Conventional therapy; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented training (TOT) (Experimental): Task-oriented training consisted of different functional tasks for lower limbs to improve balance and walk
  Interventions: Other: Task oriented training
- Conventional rehabilitation treatment (Active Comparator): Conventional rehabilitation treatment includes mat activities and range of motion (ROM) of all limbs, Lower limb strengthening and stretching, walking, cycling
  Interventions: Other: Conventional rehabilitation treatment

INTERVENTIONS:
Other: Task oriented training — Task oriented training consisted of different functional tasks for lower limbs to improve balance and walk. Each task was given 5 minutes Tasks were progressed according to each child's performance. These progressions included increase of repetitions, speed and switching between the tasks. One hour practice of these tasks was advised for home plan
  Arms: Task-oriented training (TOT)
Other: Conventional rehabilitation treatment — Conventional rehabilitation treatment includes mat activities and ROM of all limbs, Lower limb strengthening and stretching, walking, cycling.
  Each exercise was performed for 5 minutes. One hour practice of above exercises and thermotherapy for the spastic muscles advised for 10 minutes once a day at home was advised.
  Arms: Conventional rehabilitation treatment

SUMMARY:
The purpose of the study was to determine the effects of task oriented training (TOT) on walking and balance in children with spastic Cerebral Palsy (CP).

DETAILED DESCRIPTION:
The aim of study is to evaluate the effectiveness of task-oriented training on the walking in Cerebral Palsy children and compare its results with that of the conservative rehabilitation treatment. By training children to walk using task oriented training not only improves their walk and balance but also encourage them to actively participate in their own treatment process. Task oriented training approach can prove to be an effective technique for those CP children who can perform ambulation and have defined targets for gross motor activities

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP children of age between 4 to 14 years
* With spasticity 2 or less on Modified Ashworth scale
* Who can walk (GMFCS level 1-3) and can
* Can perform different activities on command

Exclusion Criteria:

* Children with cognitive impairment
* Lower limb surgery in last 6 months
* Tetraplegic CP and who are unable to walk and follow command

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test (TUG) | 6th week
  A line was marked on floor at a distance at a distance of 3 meters (9.8 feet) leveled walking. A score of 30 seconds or more suggests that the person may be prone to falls. Alternatively, a recommended practical cut-off value for the TUG to indicate normal versus below normal performance is 12 seconds.
Functional Walking Test (FWT) | 6th week
  The purpose of function walk test is to evaluate the walking balance and functional walking ability of a child. It has 5 main components. With different scores each, that is 3, 2 and 1. Also it specifies if there is any asymmetry between Right and Left lower limb and better limb functioning is recorded. Total score of FWT is 23 points
Modified Ashworth scale (MAS) | 6th week
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform.
  A score of 1 indicates no resistance, and 5 indicates rigidity.
Gross Motor Function Classification System (GMFCS) | 6th week
  GMFCS divides the CP children into 5 levels, where level 1 is the least affected and most functional children and level 5 most affected and least functional.

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Rehabilitation Medicine (AFIRM), Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toovey R, Bernie C, Harvey AR, McGinley JL, Spittle AJ. Task-specific gross motor skills training for ambulant school-aged children with cerebral palsy: a systematic review. BMJ Paediatr Open. 2017 Aug 11;1(1):e000078. doi: 10.1136/bmjpo-2017-000078. eCollection 2017. PMID 29637118
- [Background] Granild-Jensen JB, Rackauskaite G, Flachs EM, Uldall P. Predictors for early diagnosis of cerebral palsy from national registry data. Dev Med Child Neurol. 2015 Oct;57(10):931-5. doi: 10.1111/dmcn.12760. Epub 2015 Apr 9. PMID 25855100
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Pavone, V. and G. Testa, Classification of cerebral Palsy. Orthopedic Management of Children with Cerebral Palsy. A Comprehensive Approach, eds F. Canavese, and J. Deslandes (New York, NY: NOVA), 2015: p. 75-98.
- [Background] Sankar C, Mundkur N. Cerebral palsy-definition, classification, etiology and early diagnosis. Indian J Pediatr. 2005 Oct;72(10):865-8. doi: 10.1007/BF02731117. PMID 16272660
- [Background] Rethlefsen SA, Ryan DD, Kay RM. Classification systems in cerebral palsy. Orthop Clin North Am. 2010 Oct;41(4):457-67. doi: 10.1016/j.ocl.2010.06.005. PMID 20868878
- [Background] Kim, J.-H. and Y.-E. Choi, The Effect of Task-oriented Training on Mobility Function, Postural Stability in Children with Cerebral Palsy. Korean Society of Physical Medicine, 2017. 12(3): p. 79-84.
- [Background] Schiariti V, Selb M, Cieza A, O'Donnell M. International Classification of Functioning, Disability and Health Core Sets for children and youth with cerebral palsy: a consensus meeting. Dev Med Child Neurol. 2015 Feb;57(2):149-58. doi: 10.1111/dmcn.12551. Epub 2014 Aug 6. PMID 25131642
- [Background] Boyd RN, Jordan R, Pareezer L, Moodie A, Finn C, Luther B, Arnfield E, Pym A, Craven A, Beall P, Weir K, Kentish M, Wynter M, Ware R, Fahey M, Rawicki B, McKinlay L, Guzzetta A. Australian Cerebral Palsy Child Study: protocol of a prospective population based study of motor and brain development of preschool aged children with cerebral palsy. BMC Neurol. 2013 Jun 11;13:57. doi: 10.1186/1471-2377-13-57. PMID 23758951
- [Background] Paneth N. Establishing the diagnosis of cerebral palsy. Clin Obstet Gynecol. 2008 Dec;51(4):742-8. doi: 10.1097/GRF.0b013e318187081a. PMID 18981799
- [Background] Novak I, Hines M, Goldsmith S, Barclay R. Clinical prognostic messages from a systematic review on cerebral palsy. Pediatrics. 2012 Nov;130(5):e1285-312. doi: 10.1542/peds.2012-0924. Epub 2012 Oct 8. PMID 23045562
- [Background] Krigger KW. Cerebral palsy: an overview. Am Fam Physician. 2006 Jan 1;73(1):91-100. PMID 16417071
- [Background] Ketelaar M, Vermeer A, Hart H, van Petegem-van Beek E, Helders PJ. Effects of a functional therapy program on motor abilities of children with cerebral palsy. Phys Ther. 2001 Sep;81(9):1534-45. doi: 10.1093/ptj/81.9.1534. PMID 11688590
- [Background] Reid LB, Rose SE, Boyd RN. Rehabilitation and neuroplasticity in children with unilateral cerebral palsy. Nat Rev Neurol. 2015 Jul;11(7):390-400. doi: 10.1038/nrneurol.2015.97. Epub 2015 Jun 16. PMID 26077839
- [Background] Woollacott MH, Shumway-Cook A. Postural dysfunction during standing and walking in children with cerebral palsy: what are the underlying problems and what new therapies might improve balance? Neural Plast. 2005;12(2-3):211-9; discussion 263-72. doi: 10.1155/NP.2005.211. PMID 16097489
- [Background] Scrutton, D., Management of the motor disorders of children with cerebral palsy. 1984: Cambridge University Press.
- [Background] Brown, G.T. and S.A. Burns, The efficacy of neurodevelopmental treatment in paediatrics: a systematic review. British Journal of occupational therapy, 2001. 64(5): p. 235-244.
- [Background] Borggraefe I, Schaefer JS, Klaiber M, Dabrowski E, Ammann-Reiffer C, Knecht B, Berweck S, Heinen F, Meyer-Heim A. Robotic-assisted treadmill therapy improves walking and standing performance in children and adolescents with cerebral palsy. Eur J Paediatr Neurol. 2010 Nov;14(6):496-502. doi: 10.1016/j.ejpn.2010.01.002. Epub 2010 Feb 6. PMID 20138788
- [Background] McGibbon NH, Andrade CK, Widener G, Cintas HL. Effect of an equine-movement therapy program on gait, energy expenditure, and motor function in children with spastic cerebral palsy: a pilot study. Dev Med Child Neurol. 1998 Nov;40(11):754-62. doi: 10.1111/j.1469-8749.1998.tb12344.x. PMID 9881805
- [Background] Bumin G, Kayihan H. Effectiveness of two different sensory-integration programmes for children with spastic diplegic cerebral palsy. Disabil Rehabil. 2001 Jun 15;23(9):394-9. doi: 10.1080/09638280010008843. PMID 11394590
- [Background] Lim H, Kim T. Effects of vojta therapy on gait of children with spastic diplegia. J Phys Ther Sci. 2013 Dec;25(12):1605-8. doi: 10.1589/jpts.25.1605. Epub 2014 Jan 8. PMID 24409030
- [Background] Rensink M, Schuurmans M, Lindeman E, Hafsteinsdottir T. Task-oriented training in rehabilitation after stroke: systematic review. J Adv Nurs. 2009 Apr;65(4):737-54. doi: 10.1111/j.1365-2648.2008.04925.x. Epub 2009 Feb 9. PMID 19228241